CLINICAL TRIAL: NCT02582697
Title: Phase 3 Accelerated BEP: A Randomised Phase 3 Trial of Accelerated Versus Standard BEP Chemotherapy for Patients With Intermediate and Poor-risk Metastatic Germ Cell Tumours
Brief Title: Accelerated v's Standard BEP Chemotherapy for Patients With Intermediate and Poor-risk Metastatic Germ Cell Tumours
Acronym: P3BEP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Cancer Trials Ireland (Network); Children's Oncology Group (Network); Dana-Farber Cancer Institute (Other); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANZUP1302; ACTRN12613000496718 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2015-09-07; First posted 2015-10-21 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Germ Cell Tumor
Keywords: Germ Cell; Intermediate and poor-risk metastatic germ cell tumours
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Bleomycin; Injections; Etoposide; etoposide phosphate; Cisplatin; pegfilgrastim; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Arm - Standard BEP (Active Comparator): Participants 16 years or older will receive 4 cycles of Standard BEP as follows:
  * Bleomycin 30,000 IU IV weekly for 3 doses
  * Etoposide 100 mg/m2 IV on day 1 - 5
  * Cisplatin 20 mg/m2 IV on day 1 - 5
  * Pegylated G-CSF 6 mg SCI on day 6
  Patients < 16 years old and weighs ≥ 45 kg will receive:
  * Bleomycin *15,000 - 30,000 IU IV weekly for 3 doses
  * Etoposide 100 mg/m2 IV on day 1 - 5
  * Cisplatin 20 mg/m2 IV on day 1 - 5
  * Pegylated G-CSF 6 mg SCI on day 6
  Patients <16 years old and weighs < 45 kg will receive:
  * Bleomycin *15,000 - 30,000 IU IV weekly for 3 doses
  * Etoposide 100 mg/m2 IV on day 1 - 5
  * Cisplatin 20 mg/m2 IV on day 1 - 5
  * Filgrastim 10mcg/kg/day on day 6, until post-nadir Absolute Neutrophil Count ≥1 x10^9/ L
    * The dose of bleomycin is decided by the treating physician and based on the patient's Body Surface Area.
  Each cycle is 3 weeks (21 days).
  The planned total duration of treatment is 12 weeks.
  Interventions: Drug: Bleomycin (active name: Bleomycin Sulfate); Drug: Etoposide; Drug: Cisplatin; Drug: Pegylated G-CSF (Pegfilgrastim); Drug: Filgrastim
- Experimental Arm - Accelerated BEP (Experimental): Participants 16years or older will receive 4 cycles of Accelerated BEP as follows:
  * Bleomycin 30,000 IU IV wkly for 2 doses
  * Etoposide 100 mg/m2 IV on day 1 - 5
  * Cisplatin 20 mg/m2 IV on day 1- 5
  * Pegylated G-CSF 6 mg SCI on day 6
  Patients <16years and weighs ≥45 kg will receive:
  * Bleomycin *15,000 - 30,000 IU IV wkly for 2 doses
  * Etoposide 100 mg/m2 IV on day 1 - 5
  * Cisplatin 20 mg/m2 IV on day 1 - 5
  * Pegylated G-CSF 6 mg SCI on day 6
  Patients <16years and weighs <45 kg will receive:
  * Bleomycin *15,000 - 30,000 IU IV wkly for 2 doses
  * Etoposide 100 mg/m2 IV on day 1 - 5
  * Cisplatin 20 mg/m2 IV on day 1 - 5
  * Filgrastim 10mcg/kg/day on day 6, until ANC ≥1 x10^9/ L
  Each cycle is 2 weeks (14days)
  Following 4xBEP cycles, patients will receive additional bleomycin as follows:
  - Bleomycin *15,000 - 30,000 IU IV wkly for 4 doses
  * The dose of bleomycin is decided by the treating physician and based on the patient's BSA.
  The planned total duration is 12 weeks.
  Interventions: Drug: Bleomycin (active name: Bleomycin Sulfate); Drug: Etoposide; Drug: Cisplatin; Drug: Pegylated G-CSF (Pegfilgrastim); Drug: Filgrastim

INTERVENTIONS:
Drug: Bleomycin (active name: Bleomycin Sulfate) — Standard Arm: Bleomycin 30,000 international units IV weekly for 3 doses (eg. days 1, 8 and 15 or days 2, 9 and 16 of a 21-day cycle) for 4 cycles.
  Accelerated Arm: Bleomycin 30,000 international units IV weekly for 2 doses (eg. days 1 and 8 or days 2 and 9 of a 14-day cycle) for 4 cycles. Followed by Bleomycin 30,000 international units IV weekly for 4 doses.
  Other Names: Blenamax (Aspen); DBL Bleomycin Sulphate (Willow Pharmaceuticals Pty Limited); Bleo Powder for injection (Hospira)
Drug: Etoposide — Standard Arm: Etoposide 100 mg/m2 IV on days 1, 2, 3, 4, 5 of a 21-day cycle for 4 cycles.
  Accelerated Arm: 100 mg/m2 IV on days 1, 2, 3, 4, 5 of a 14-day cycle for 4 cycles.
  Other Names: DBL Etoposide Injection (Hospira); Etopophos (Bristol-Myers Squibb); Etoposide (Pfizer); Etoposide Ebewe (Sandoz)
Drug: Cisplatin — Standard Arm: Cisplatin 20 mg/m2 IV on days 1, 2, 3, 4, 5 of a 21-day cycle for 4 cycles.
  Accelerated Arm: Cisplatin 20 mg/m2 IV on days 1, 2, 3, 4, 5 of a 14-day cycle for 4 cycles.
  Other Names: Cisplatin Ebewe (Sandoz); Cisplatin injection (Pfizer); DBL Cisplatin Injection (Hospira)
Drug: Pegylated G-CSF (Pegfilgrastim) — Standard Arm: 6 mg SCI on day 6 of a 21-day cycle for 4 cycles. Accelerated Arm: 6 mg SCI on day 6 of a 14-day cycle for 4 cycles.
  Other Names: Neulasta Syringe with Automatic Needle Guard (Amgen)
Drug: Filgrastim — Standard Arm: 10 mcg/kg/day on day6, until post-nadir absolute neutrophil count ≥ 1.0 x 10^9/L, of a 21-day cycle for 4 cycles.
  Accelerated Arm: 10 mcg/kg/day on day 6, until post-nadir absolute neutrophil count ≥ 1.0 x 10^9/L, of a 14-day cycle for 4 cycles.
  Other Names: Neupogen (Amgen); Nivestim (Hospira); Tevagrastim (Teva Pharma Australia Pty Ltd); Zarzio (Sandoz)

SUMMARY:
The purpose of this study is to determine whether accelerated BEP chemotherapy is more effective than standard BEP chemotherapy in males with intermediate and poor-risk metastatic germ cell tumours.

DETAILED DESCRIPTION:
Bleomycin, Etoposide, Cisplatin (BEP) administered 3-weekly x 4 remains standard 1st line chemotherapy for intermediate- and poor-risk metastatic germ cell tumours (GCTs). Cure rates are over 90% for good-risk disease, 85% with intermediate-risk, and about 70% for poor-risk disease. Previous strategies to improve first-line chemotherapy have failed to improve cure rates and were more toxic than BEP. New strategies are needed for patients with intermediate and poor-risk disease. BEP is accelerated by cycling Cisplatin and etoposide 2-weekly instead of 3-weekly. The Australian and New Zealand Urogenital and Prostate Cancer Trials Group (ANZUP) is conducting a trial comparing accelerated BEP with standard BEP. The aim of this study is to determine if accelerated BEP is superior to standard BEP as first-line chemotherapy for intermediate and poor risk metastatic GCTs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 11 years and ≤ 50 years on the date of randomisation
2. Histologically or cytologically confirmed germ cell tumour (non-seminoma or seminoma); or Exceptionally raised tumour markers (AFP ≥ 1000ng/mL and/or HCG ≥ 5000 IU/L) without histologic or cytologic confirmation in the rare case where pattern of metastases consistent with GCT, high tumour burden, and a need to start therapy urgently
3. Primary arising in testis, ovary, retro-peritoneum, or mediastinum
4. Metastatic disease or non-testicular primary
5. Intermediate or poor prognosis as defined by IGCCC classification3 (modified with different LDH criteria for intermediate risk non-seminoma, and inclusion of ovarian primaries). (See protocol for more information).
6. Adequate bone marrow function with ANC ≥1.0 x 10^9/L, Platelet count ≥100 x 10^9/L
7. Adequate liver function where bilirubin must be ≤1.5 x ULN, except participants with Gilbert's Syndrome where bilirubin must be ≤2.0 x ULN; ALT and AST must be ≤2.5 x ULN, except if the elevations are due to hepatic metastases, in which case ALT and AST must be ≤ 5 x ULN
8. Adequate renal function with estimated creatinine clearance of ≥60 ml/min according to the Cockcroft-Gault formula, unless calculated to be < 60 ml/min or borderline in which case GFR should be formally measured, eg. with EDTA scan
9. ECOG Performance Status of 0, 1, 2, or 3
10. Study treatment both planned and able to start within 14 days of randomisation.
11. Willing and able to comply with all study requirements, including treatment, timing and nature of required assessments
12. Able to provide signed, written informed consent

Exclusion Criteria:

1. Other primary malignancy (EXCEPT adequately treated non-melanomatous carcinoma of the skin, germ cell tumour, or other malignancy treated at least 5 years previously with no evidence of recurrence)
2. Previous chemotherapy or radiotherapy, except if patient has pure seminoma relapsing after adjuvant radiotherapy or adjuvant chemotherapy with 1-2 doses of single agent carboplatin or if patient hasb. non-seminoma by IGCCC criteria or stage IV malignant ovarian germ cell tumour in the rare case where low-dose induction chemotherapy is given prior to registration because patient is not fit enough to receive protocol chemotherapy (eg. organ failure, vena cava obstruction, overwhelming burden of disease). Acceptable regimens include cisplatin 20 mg/m2 days 1-2 and etoposide 100 mg/m2 days 1-2; carboplatin AUC 3 days 1-2 and etoposide 100 mg/m2 days 1-2; or baby-BOP.43 Patients must meet all other inclusion and exclusion criteria at the time of registration.

   Additionally participants who need to start therapy urgently prior to completing study-specific baseline investigations may commence study chemotherapy prior to registration and randomisation. Such patients must be discussed with the coordinating centre prior to registration, and must be registered within 10 days of commencing study chemotherapy.
3. Significant cardiac disease resulting in inability to tolerate IV fluid hydration for cisplatin
4. Significant co-morbid respiratory disease that contraindicates the use of bleomycin
5. Peripheral neuropathy ≥ grade 2 or clinically significant sensorineural hearing loss or tinnitus
6. Concurrent illness, including severe infection that may jeopardize the ability of the participant to undergo the procedures outlined in this protocol with reasonable safety
7. Inadequate contraception. Men must use 2 effective methods of contraception, including use of a condom, during chemotherapy and for a year after completing chemotherapy.
8. Known allergy or hypersensitivity to any of the study drugs
9. Presence of any psychological, familial, sociological or geographical condition that in the opinion of the investigator would hamper compliance with the study protocol and follow-up schedule, including alcohol dependence or drug abuse

The above inclusion and exclusion criteria will apply to stage 1 (n=150) and stage 2 (n=500 including stage 1) of the study. All sites will participate in both stages of the study with the exception of the Children's Oncology Group who will be participate in stage 1 only.

Ages: 11 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (disease progression or death) | From randomisation up to disease progression or date of death whichever come first, assessed up to 5 years
  PFS is measured from the date of randomisation until the criteria for disease progression are met (as defined in the protocol) or death. Participants who are not observed to progress nor die will be censored at the date of last follow-up

SECONDARY OUTCOMES:
Initial response assessment | At end of chemotherapy treatment, treatment planned for 12 weeks
  The assessment of response of germ cell tumours is measured by the change in size of measurable tumour masses in combination with changes in serum tumour markers after chemotherapy treatment.
Final response assessment | At 6 months
  The assessment of response of germ cell tumours is measured by changes in serum tumour markers and imaging at 6 months from randomisation, or after any post-chemotherapy surgical resection or other intervention, whichever occurs last.
Adverse events (worst grade according to NCI CTCAE v4.03) | From start of chemotherapy until 30 days after last dose, an average of 4 months
  The intensity of adverse events will be assessed using the NCI Common Terminology Criteria for Adverse Events version 4 (NCI CTCAE v4.03)
Health-related quality of life | From date of randomisation until date of 18 month follow-up
  HR-QoL measures will include the EORTC core quality of life questionnaire (QLQ-C30), a 30-item cancer-specific questionnaire that is well-validated and available in many languages.
Health-related quality of life for testicular cancer | From date of randomisation until date of 18 month follow-up
  EORTC quality of life module for testicular cancer (QLQ-TC26), a disease-specific measure with 26 items about physical symptoms, sexual functioning and emotional issues.
Treatment preference | From date of randomisation until date of 18 month follow-up
  A trial-specific preferences question will be used to determine if participants think they would prefer to be treated with accelerated BEP or standard BEP, assuming that they were equally effective.
Delivered dose-intensity of chemotherapy (relative to standard BEP) | From start date of chemotherapy treatment until date of end of chemotherapy, an average of 12 weeks
  Delivered dose-intensity of cisplatin, etoposide and bleomycin will be assessed.
Overall survival | From randomisation up to disease progression or date of death whichever come first, assessed up to 5 years
  Overall survival is measured from the date of randomisation until death from any cause, or the date of last known follow-up alive.

OTHER OUTCOMES:
Exploratory biomarker investigations | Baseline
  Associations between biomarkers with survival will be assessed in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Grimison, Study Chair — Chris O'Brien Lifehouse
Locations (28):
- Memorial Sloan Kettering Cancer Centre, New York, New York, United States
- Australia (22):
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Chris O'Brien Lifehouse, Sydney, New South Wales
  - Macquarie Cancer Clinical Trials, Sydney, New South Wales
  - Concord Repatriation General Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Nepean Hospital, Sydney, New South Wales
  - Tweed Hospital, Tweed Heads, New South Wales
  - SAN Clinical Trials Unit, Wahroonga, New South Wales
  - Royal Brisbane & Women's Hospital, Brisbane, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Princess Alexandra, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Austin Health, Heidelberg, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- New Zealand (5):
  - Starship Children's Hospital, Grafton, Auckland
  - Auckland Hospital, Grafton, Auckland
  - Palmerston North Hospital, Roslyn, Palmerston North
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin

REFERENCES:
- [Derived] Lawrence NJ, Chan H, Toner G, Stockler MR, Martin A, Yip S, Wong N, Yeung A, Mazhar D, Pashankar F, Frazier L, McDermott R, Walker R, Tan H, Davis ID, Grimison P; ANZUP. Protocol for the P3BEP trial (ANZUP 1302): an international randomised phase 3 trial of accelerated versus standard BEP chemotherapy for adult and paediatric male and female patients with intermediate and poor-risk metastatic germ cell tumours. BMC Cancer. 2018 Aug 29;18(1):854. doi: 10.1186/s12885-018-4745-3. PMID 30157803